CLINICAL TRIAL: NCT03286270
Title: A mRUS Validation Study for Nail-treated Fractures of Long Bones and a TUS Exploratory Study for Nail and Plate-treated Fractures of Long Bones
Acronym: mRUSTUS
Status: Completed | Type: Observational
Sponsor: Bone Therapeutics S.A (Industry)
Responsible Party: Sponsor
Other Study IDs: 002A/BT
Record Dates: First submitted 2017-09-15; First posted 2017-09-18 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Delayed Union Fracture; CT-scan; X-Ray; Bone Fracture; Fracture Healing; Validation Studies
Keywords: mRUS; validation tool; Impaired fractures
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early intervention attempts to shorten protracted delayed union (DU) or prevent non-union (NU) fractures are hampered by lack of validated quantitative assessment tools for bone fracture healing during normal and delayed healing processes. In actual practice, sequential X-rays usually follow a pre-determined time interval in patients with fractures.They constitute the best available state of the art used by surgeons to assess the fracture healing course.

In an attempt to improve between raters reliability of radiographic assessment of healing, studies have explored a novel radiographic assessment for tibial shaft fractures, the Radiographic Union Scale for Tibial Fractures (RUST). The RUST assesses the presence of bridging callus and a fracture line on each of four cortices (seen on anterior-posterior and lateral views). This callus based scoring system has been since extended to other bones than the tibia in a retrospective case series. It has been renamed modified radiological union score (mRUS) and has shown potential value in bone healing measurement.

Based on an initial retrospective study in nail-treated fractures, the first objective of the present investigation is to prospectively validate mRUS as a tool to identify patients at increased risk of DU and NU within the first 75-110 days after fracture occurrence. This prospective validation will be performed on a retrospective cohort of patients having sustained long bone fractures, including both upper and lower extremities. A further objective of the present investigation is to apply the scoring system to tomographic imaging in case of nail/plate treated fractures, deriving a tomographic union score (TUS) and first assess its potential value in bone healing for fractures treated by nails/plates.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patient (>18 and < 80 years old)
* Patient with nail(s) (for mRUS validation study and TUS exploratory study) or plate(s) (for TUS exploratory study) treated long bone fractures, corresponding to the following OA/OTA classification: 11-A, 12-A, -B and -C, 13-A, 21-A, 22-A, -B and -C, , 31-A3, 32-A, -B and -C, 33-A 41-A2 and A3, 42-A, -B and -C and 43-A
* Patient for whom outcome of fracture is known
* For the mRUS validation study, patient with one follow up X-ray imaging performed 75-110 days after fracture occurrence
* For the TUS exploratory study, patient with one follow up CT-scan imaging performed 75-110 days after the fracture occurrence

Exclusion Criteria:

* Bone infection diagnosed between time of the fracture occurrence and the X-Ray or CT-scan imaging performed 75-110 days after the fracture occurrence
* Previous fracture and previous surgery on the fractured bone
* Bone tumour or history of bone tumour
* Bone metastasis
* Known evidence for ongoing metabolic bone disease (e.g. chronic renal failure, hyper or hypoparathyroidism, rickets, Paget's disease of bone, inherited or congenital bone abnormalities)
* Patient with current traumatic brain injury

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Long bone fracture
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
mRUS assessed on X-Ray | 75-110 days after fracture occurrence

SECONDARY OUTCOMES:
TUS assessed on CT-scan | 75-110 days after fracture occurrence

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Investigating site DE01, Cologne
  - Investigating site DE03, Lübeck
  - Investigating site DE02, Munich
  - Investigating site DE04, Würzburg